CLINICAL TRIAL: NCT02702115
Title: A Phase I / 2, Multicenter, Open-label, Single-dose, Dose-ranging Study to Assess the Safety and Tolerability of SB-318, a rAAV2/6-based Gene Transfer in Subjects With Mucopolysaccharidosis I (MPS I)
Brief Title: Ascending Dose Study of Genome Editing by the Zinc Finger Nuclease (ZFN) Therapeutic SB-318 in Subjects With MPS I
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: All three subjects dosed in the study have rolled over to the Long-Term Follow-up Study IVPRP-LT01 (NCT04628871)
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-318-1502
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-12

CONDITIONS: MPS I
Keywords: Mucopolysaccharidosis I; MPS I; Hurler-Scheie syndrome; Gene Therapy; Gene Editing; Zinc Finger; SB-318; Rare; Genetic; DNA; Sangamo; Genome editing; Empowers; ZFN; Hurler; Gene Specific Targeted Insertion
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: SB-318: Starting Dose 1.00E+13 vg/kg (Experimental): A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-318
- Cohort 2: SB-318 at Next Ascending Dose 5.00E+13 vg/kg (Experimental): A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-318
- Cohort 3: SB-318 at Next Ascending Dose 1.20E+14 vg/kg (Experimental): A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  Interventions: Biological: SB-318

INTERVENTIONS:
Biological: SB-318 — A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability of ascending doses of SB-318. SB-318 is an intravenously delivered Zinc Finger Nuclease (ZFN) Therapeutic for genome editing. It inserts a correct copy of the α-L-iduronidase (IDUA) gene into the Albumin locus in hepatocytes with the goal of lifelong therapeutic production of the IDUA enzyme.

DETAILED DESCRIPTION:
The objectives of the study are to provide long term expression of IDUA and improve the current clinical outcome of enzyme replacement therapy (ERT) or hematopoietic stem cell transplantation (HSCT) therapy in subjects with attenuated MPS I, a recessive lysosomal storage disorder that results from mutations in the gene encoding IDUA. SB-318 is a therapeutic for ZFN-mediated genome editing which will be delivered by adeno-associated virus (AAV)-derived vectors. SB-318 is intended to function by placement of the corrective copy of the IDUA transgene into the genome of the subject's own hepatocytes, under the control of the highly expressed endogenous albumin locus, and is expected to provide permanent, liver-specific expression of iduronidase for the lifetime of an MPS I patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 5 years of age
* Clinical diagnosis of attenuated MPS I deficiency (Hurler-Scheie, Scheie, or Hurlers status post-HSCT)

Exclusion Criteria:

* Known to be unresponsive to ERT
* Neutralizing antibodies to AAV 2/6
* Serious intercurrent illness or clinically significant organic disease (unless secondary to MPS I)
* Receiving antiviral therapy for hepatitis B or C, or with active hepatitis B or hepatitis C or HIV 1/2
* Lack of tolerance to laronidase treatment with significant IARs or occurrence of anaphylaxis
* Markers of hepatic dysfunction
* Creatinine ≥ 1.5 mg/dL
* Contraindication to the use of corticosteroids for immunosuppression
* Current treatment with systemic (IV or oral) immunomodulatory agent or steroid use (topical treatment allowed)
* Participation in prior investigational drug or medical device study within the previous 3 months
* Prior treatment with a gene therapy product
* Elevated or abnormal circulating α-fetoprotein (AFP)
* Weight <20 kg at Screening Visit

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

REFERENCES:
- [Derived] Harmatz P, Prada CE, Burton BK, Lau H, Kessler CM, Cao L, Falaleeva M, Villegas AG, Zeitler J, Meyer K, Miller W, Wong Po Foo C, Vaidya S, Swenson W, Shiue LH, Rouy D, Muenzer J. First-in-human in vivo genome editing via AAV-zinc-finger nucleases for mucopolysaccharidosis I/II and hemophilia B. Mol Ther. 2022 Dec 7;30(12):3587-3600. doi: 10.1016/j.ymthe.2022.10.010. Epub 2022 Oct 25. PMID 36299240
- [Derived] Ou L, Przybilla MJ, Ahlat O, Kim S, Overn P, Jarnes J, O'Sullivan MG, Whitley CB. A Highly Efficacious PS Gene Editing System Corrects Metabolic and Neurological Complications of Mucopolysaccharidosis Type I. Mol Ther. 2020 Jun 3;28(6):1442-1454. doi: 10.1016/j.ymthe.2020.03.018. Epub 2020 Apr 8. PMID 32278382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original protocol anticipated 9-12 subjects in 3 cohorts at ascending doses. However, enrollment ended after 3 subjects were enrolled in 2 cohorts. (No subjects were enrolled in cohort 3). After interim data analysis, the sponsor decided to stop enrollment in this study at 3 subjects enrolled, all adults, in 2 cohorts. (No subjects were enrolled in cohort 3) The sponsor continues to monitor the subjects in a 10-year,follow-up study ST-IVPRP-LT01 (NCT04628871).
Groups:
- Cohort 1: SB-318: Starting Dose 1.00E+13vg/kg: A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
- Cohort 2: SB-318 at Next Ascending Dose 5.00E+13vg/kg; Cohort 3: SB-318 at Next Ascending Dose 1.20E+14vg/kg: A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
  SB-318: A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
Period: Overall Study
Arm/Group | Cohort 1: SB-318: Starting Dose 1.00E+13vg/kg | Cohort 2: SB-318 at Next Ascending Dose 5.00E+13vg/kg | Cohort 3: SB-318 at Next Ascending Dose 1.20E+14vg/kg
Started | 1 | 2 | 0
Completed | 1 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The original protocol anticipated 9-12 subjects in 3 cohorts at ascending doses. However, enrollment ended after 3 subjects were enrolled in 2 cohorts. (No subjects were enrolled in cohort 3). After interim data analysis, the sponsor decided to stop enrollment in this study at 3 subjects enrolled, all adults, in 2 cohorts. (No subjects were enrolled in cohort 3) The sponsor continues to monitor the subjects in a 10-year,follow-up study ST-IVPRP-LT01 (NCT04628871).
Groups:
- Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg; Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg; Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg: SB-318: A single dose of each of the three components of SB-318 [zinc finger nucleases (ZFN1, ZFN2, and hIDUA Donor)] administered via intravenous (IV) infusion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg | Total
Number analyzed (Participants) | 1 | 2 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 0 | 3
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 |  | 3
Baseline Iduronidase (IDUA) Activity [Mean (Standard Deviation); unit: nmol/hr/mg] | 1.200 (NA) — There was only one subject in this cohort | 9.955 (2.7789) |  | 7.037 (5.4232)
Baseline Urine Glycosaminoglycans (GAG Levels) [Mean (Standard Deviation); unit: g/mol creatinine]
  Dermatan Sulfate, Urine | 129.3500 (NA) — There was only one subject in this cohort | 15.6680 (6.37527) |  | 53.5620 (65.78896)
  Heparan Sulfate Urine | 109.4200 (NA) — There was only one subject in this cohort | 12.3345 (3.72575) |  | 44.6963 (56.11422)
  Total GAG | 11.360 (NA) — There was only one subject in this cohort | 3.620 (0.8485) |  | 6.200 (4.5088)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of Participants with Treatment-Emergent Adverse Events
Time Frame: Up to 36 months after the SB-318 infusion
Population: No subjects were enrolled in Cohort 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg
Number analyzed (Participants) | 1 | 2 | 0
Participants | 1 | 2 | 0

2. Secondary Outcome: Effect of SB-318 on IDUA Activity
Description: Change from baseline clinical laboratory in measurement of IDUA activity measured in leukocytes.
Time Frame: Baseline and Month 36 after the SB-318 infusion
Population: No subjects were enrolled in Cohort 3
Measure: Mean (Standard Deviation); unit: nmol/hr/mg
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg
Number analyzed (Participants) | 1 | 2 | 0
nmol/hr/mg | -1.200 (NA) — Only one subject was enrolled in Cohort 1 | -2.515 (5.9185) |

3. Secondary Outcome: Effect of SB-318 on Urine Glycosaminoglycans (GAG) Levels
Description: Change from baseline in total GAG, Dermatan Sulfate GAG, and Heparan Sulfate GAG measured in urine at Month 24
Time Frame: Baseline and 24 months after the SB-318 infusion
Population: No subjects were enrolled in Cohort 3
Measure: Mean (Standard Deviation); unit: g/mol creatinine
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg
Number analyzed (Participants) | 1 | 2 | 0
g/mol creatinine
  Dermatan Sulfate | 0.510 (NA) — Only one subject was enrolled in Cohort 1 | -0.090 (0.3960) |
  Heparan Sulfate | 30.2000 (NA) — Only one subject was enrolled in Cohort 1 | 3.6005 (8.22436) |
  Total GAG | 0.940 (NA) — Only one subject was enrolled in Cohort 1 | 0.240 (0.0424) |

4. Secondary Outcome: AAV2/6 Clearance in Plasma, Saliva, Urine, Stool, and Semen
Description: Subjects with AAV2/6 clearance in plasma, saliva, urine, stool, and semen by PCR by Week 24.
Time Frame: Up to 24 months after the SB-318 infusion
Population: No subjects were enrolled in Cohort 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg
Number analyzed (Participants) | 1 | 2 | 0
Participants | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the subject's date of screening until their end of study visit at 36 months.
Description: No subjects were enrolled in Cohort 3
Arm/Group | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg (N=1) | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg (N=2) | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg (N=0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | NA
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | NA
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | NA
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1: SB-318: Starting Dose_1.00E+13 vg/kg (N=1) | Cohort 2: SB-318 at Next Ascending Dose_5.00E+13 vg/kg (N=2) | Cohort 3: SB-318 at Next Ascending Dose_1.20E+14 vg/kg (N=0)
Aortic valve stenosis (Cardiac disorders) | 0/0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0/0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | NA
Left atrial enlargement (Cardiac disorders) | 1 (1) | 0 (0) | NA
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | NA
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | NA
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | NA
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Blood cortisol decreased (Investigations) | 0 (0) | 2 (2) | NA
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | NA
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | NA
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | NA
Upper Respiratory Infection (Infections and infestations) | 1 (2) | 2 (4) | NA
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA
Headache (Nervous system disorders) | 1 (2) | 1 (2) | NA
Renal Cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Continuous data will be summarized using the following descriptive statistics: the number of subjects (n), mean, standard deviation (SD), median, minimum and maximum, where appropriate. Categorial percentage (%) of subjects for each category, where appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT02702115/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02702115/SAP_001.pdf